CLINICAL TRIAL: NCT02192034
Title: Optimizing Navigation to Successful Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: ACS255086
Record Dates: First submitted 2014-06-02; First posted 2014-07-16 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer Screening
Keywords: Colonoscopy; Colon cancer; screening; navigation
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navigation Group (Experimental): This group will receive standard clinic instructions for the colonoscopy and two additional phone calls from the patient navigator to discuss the purpose, preparation, and additional information regarding the colonoscopy procedure.
  Interventions: Behavioral: Navigation
- Control (Placebo Comparator): This group will receive only clinic instructions without intervention from the patient navigator.
  Interventions: Behavioral: Navigation

INTERVENTIONS:
Behavioral: Navigation

SUMMARY:
Colorectal cancer is the second leading cause of death from cancer in the United States. Two major barriers to successful colorectal cancer screening are appointment keeping and proper bowel preparation. The purpose of this study is to test the efficacy of a patient navigation program to increase colorectal cancer screening at Rush University Medical Center. The investigators hypothesize that colorectal cancer screening will be improved for subjects who utilize a patient navigator.

ELIGIBILITY:
Inclusion Criteria:

* Subject deemed appropriate for colorectal cancer screening by colonoscopy by a primary care physician
* Age 50 or greater or 40 or greater with family history of colorectal cancer in first degree relative
* Average risk for screening as defined as absence of symptomatic abdominal pain and active GI bleeding

Exclusion Criteria:

* Age > 75 years old
* Congestive Heart Failure
* Chronic Obstructive Pulmonary Disease
* Myocardial Infarction
* Weight greater than 350 pounds
* Anticoagulation
* Inability to speak English

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Navigation role in colorectal cancer screening | Up to 90 days
  Primary endpoint will be the role of navigation to obtain colonoscopy attendance with adequate colonoscopy preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua E Melson, MD, MPH, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States